CLINICAL TRIAL: NCT05916014
Title: Artificial Intelligence-assisted White Light Endoscopy to Identify the Kimura-Takemoto Classification of Atrophic Gastritis to Achieve Gastric Cancer Risk Assessment
Brief Title: AI-assisted White Light Endoscopy to Identify the Kimura-Takemoto Classification of Atrophic Gastritis
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Linyi County People's Hospital,Dezhou,China (Unknown)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022SDU-QILU-123
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Atrophic Gastritis; Artificial Intelligence; Endoscopy
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic atrophic gastritis observed by white light endoscope: Get pictures from gastric antrum,gastric angle,lesser curvature of gastric body, cardia, gastric fundus, greater curvature of gastric body by white light endoscope
  Interventions: Diagnostic Test: Diagnostic Test: The diagnosis of Artificial Intelligence and endosopists

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: The diagnosis of Artificial Intelligence and endosopists — Endosopists and AI will assess the Kimura-Takemoto classification independently when the patients is eligible.

SUMMARY:
Grading endoscopic atrophy according to the Kimura-Takemoto classification can assess the risk of gastric neoplasia development. However, the false negative rate of chronic atrophic gastritis is high due to the varying diagnostic standardization and diagnostic experience and levels of endoscopists. Therefore, this study aims to develop an AI model to identify the Kimura-Takemoto classification.

DETAILED DESCRIPTION:
Grading endoscopic atrophy according to the Kimura-Takemoto classification can assess the risk of gastric neoplasia development. The higher the score, the more severe the degree of atrophic gastritis. However, the false negative rate of chronic atrophic gastritis is high due to the varying diagnostic standardization and diagnostic experience and levels of endoscopists. Therefore, this study aims to develop an AI model to identify the Kimura-Takemoto classification of atrophic gastritis to achieve gastric cancer risk assessment.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-80 years who undergo the white light endoscope examination Informed consent form provided by the patient.

Exclusion Criteria:

1. patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric;
2. disorders who cannot participate in gastroscopy;
3. Patients with progressive gastric cancer;
4. low quality pictures;
5. patients with previous surgical procedures on the stomach or esophageal;
6. patients who refuse to sign the informed consent form;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the gastrointestinal endoscopy examination and screened that fulfill the eligibility criteria at Qilu Hospital,Shandong University,Linyi County People's Hospital will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI model to diagnose the Kimura-Takemoto classification | 2 years
  Accuracy of AI model to diagnose the Kimura-Takemoto classification
Sensitivity of AI model to diagnose the Kimura-Takemoto classification | 2 years
  Sensitivity of AI model to diagnose the Kimura-Takemoto classification
Specificity of AI model to diagnose the Kimura-Takemoto classification | 2 years
  Specificity of AI model to diagnose the Kimura-Takemoto classification

SECONDARY OUTCOMES:
The MIOU value of AI model in semantic segmentation of endoscopic atrophy picture | 2 years
  The MIOU value of AI model in semantic segmentation of endoscopic atrophy picture

CONTACTS AND LOCATIONS:
Overall Officials: yanqing li, MD,PHD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastrology, QiLu Hospital, Shandong University, Shangdong, Shandong, China